CLINICAL TRIAL: NCT02926092
Title: A Prospective, Multicenter, Longitudinal, Observational Natural History Study to Evaluate Disease Progression in Subjects With Autosomal Dominant Retinitis Pigmentosa (adRP) With Misfolded Rod Opsin Mutations
Brief Title: Observational Natural History Study of Autosomal Dominant Retinitis Pigmentosa (adRP)
Status: Terminated | Type: Observational
Why Stopped: Development of SHP630 was discontinued based on lack of preclinical efficacy.
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Other Study IDs: SHP630-001
Record Dates: First submitted 2016-10-05; First posted 2016-10-06 (Estimated); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Retinitis Pigmentosa
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood will be obtained during the pre-screening period
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Arm 1: Observation of progression of disease over time.
  Interventions: Diagnostic Test: Observation

INTERVENTIONS:
Diagnostic Test: Observation — Observation of progression of disease over time

SUMMARY:
The purpose of this study is to gain an understanding of how adRP progresses over time in patients with misfolded rod opsin mutations.

ELIGIBILITY:
Inclusion Criteria:

1. The subject has 1 documented pre-specified heterozygous rhodopsin gene (RHO) mutation confirmed by genetic testing (mutations will include P23H, T17M, and R135W).
2. The subject has at least 1 eye that meets all 3 of the following criteria:

   1. A measurable EZ area as determined by an evaluation of EZ limits on sdOCT scan, with a horizontal EZ width of greater than 3 mm
   2. BCVA of greater than or equal to 35 letters as measured by the Early Treatment Diabetic Retinopathy Study (ETDRS; equivalent to 20/200 on a Snellen chart).
   3. A kinetic VF of greater than 10 degrees diameter in the horizontal meridian with a spot size of III
3. The subject has the ability to comply with the clinical protocol, in the opinion of the investigator.
4. The subject has a clear ocular media and adequate pupillary dilation in both eyes to permit adequate visual assessments in the opinion of the investigator.
5. The subject has agreed to abstain from any protocol-prohibited medication(s) during study participation.
6. The subject is medically stable in the opinion of the investigator and able to fulfill the protocol requirements, including the ability to complete the assessments, without placing an undue burden on the subject/subject's family.
7. The subject and/or subject's parent(s) or legally authorized guardian(s) has voluntarily signed an Institutional Review Board (IRB)/ ethics committee (EC)-approved informed consent and assent form(s), as applicable, after all relevant aspects of the study have been explained and discussed with the subject and/or the subject's parent(s) or legally authorized guardian(s).
8. The subject, subject's parent(s), or legally authorized guardian(s) is able to understand the nature, scope, and possible consequences of the study and agrees to comply with the protocol-defined, scheduled assessments.

Exclusion Criteria:

1. The subject is participating in an interventional clinical trial or has participated in an interventional clinical trial within 90 days of screening; participation in non-interventional observational studies is permitted.
2. The subject has received treatment or has been in the treatment arm of a clinical trial for gene therapy, stem cell therapy, retinal progenitor cell therapy, tissue transplantation, device or drug delivery implantation, or other similar invasive therapy.
3. The subject has any of the following medical conditions that will interfere with consistent follow-up over any part of the study:

   1. Stroke
   2. Severe or unstable coronary disease
   3. End-stage or aggressive malignancy
   4. General poor health or uncontrolled or severe disease (eg, cardiovascular, neurological, psychological, pulmonary,renal, hepatic, endocrine, or gastrointestinal disorders) that in the opinion of the investigator would interfere with participation in the study
4. The subject has any of the following ocular conditions that could interfere with or confound follow-up of disease progression:

   * Glaucoma
   * Diabetic retinopathy
   * Choroidal neovascularization
   * Retinal inflammatory disease
   * Cataract worse than grade 2 (nuclear, posterior subcapsular [PSC], or cortical)
   * High myopia (≥8 diopters)
   * Herpes simplex virus of the eye
   * Acute infection or inflammation
   * Any ocular condition that in the opinion of the investigator would interfere with the ability to assess retinal morphology and functionality
5. The subject has had intraocular surgery within 90 days prior to screening.
6. The subject currently requires the following protocol prohibited medications or has ingested such medication within 30 days of screening:

   Plaquenil Thioridazine Clofazimine Deferoxamine Phenothiazine Chlorpromazine Cisplatin Valproic acid Any other drugs with known visual side effects
7. The subject has 3 first- or second-degree family members already enrolled in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study population will come from a clinical setting where a diagnosis of adRP has been made
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2017-03-13 (Actual); Primary Completion 2017-04-13 (Actual); Study Completion 2017-04-13 (Actual)

PRIMARY OUTCOMES:
Progression of disease over time in adRP patients with misfolded rod opsin mutations using ellipsoid zone (EZ) area measurements | Baseline to 4 years

SECONDARY OUTCOMES:
Progression of disease over time in adRP patients with misfolded rod opsin mutations as measured by EZ width | Baseline to 4 years
Progression of disease over time in adRP patients with misfolded rod opsin mutations as measured by visual fields (kinetic and static) | Baseline to 4 years
Progression of disease over time in adRP patients with misfolded rod opsin mutations as measured by dark-adapted rod visual fields | Baseline to 4 years
Progression of disease over time in adRP patients with misfolded rod opsin mutations as measured by electroretinography (ERG): dark- and light-adapted | Baseline to 4 years
Progression of disease over time in adRP patients with misfolded rod opsin mutations as measured by best corrected visual acuity (BCVA) | Baseline to 4 years
Vision-related function and quality of life as measured by 25-item National Eye Institute Visual Function Questionnaire (NEI VFQ-25) plus its additional items | Baseline to 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Shire Director, Study Director — Takeda
Locations (1):
- Texas Retina Associates,, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data from this particular study will not be shared as there is a reasonable likelihood that individual patients could be re-identified (due to the limited number of study participants).

REFERENCES:
- See also: To obtain more information on the study, click here/on this link. — https://clinicaltrials.takeda.com/study-detail/5f6b5fd94db2bf003ab47096